CLINICAL TRIAL: NCT05871697
Title: The Relationship Between Multifidus and Gastrocnemius Muscle Thickness With Postural Stability in Patients With Spinal Cord Injury
Brief Title: Multifidus & Gastrocnemius Muscle Thickness & Postural Stability in Spinal Cord Injury Patients: A Correlational Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Uskudar State Hospital (Other Government)
Collaborators: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Mustafa Hüseyin Temel, Principal Investigator, Uskudar State Hospital
Other Study IDs: SKLPosture1
Record Dates: First submitted 2023-05-08; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with spinal cord injury: Patients who have spinal cord injury.
  Interventions: Other: Measurement of multifidus and gastrocnemius muscle thickness with Ultrasound; Other: Berg Balance Scale

INTERVENTIONS:
Other: Measurement of multifidus and gastrocnemius muscle thickness with Ultrasound — To measure multifidus and gastrocnemius muscle thickness using ultrasound imaging, the following steps are typically followed. First, the patient is positioned appropriately to allow access to the muscles to be imaged. For example, the patient may lie prone for imaging of the lumbar multifidus or sit with the leg extended for imaging of the gastrocnemius. Next, a trained clinician or technician places an ultrasound probe on the skin over the target muscle and adjusts the settings on the ultrasound machine to optimize the image quality. The probe is then moved around to obtain different views of the muscle, and the images are stored for later analysis. To measure muscle thickness, the clinician or technician identifies the muscle fascia on the ultrasound image and measures the distance between the fascia and the underlying bone or tissue. This measurement provides an estimate of the muscle thickness.
Other: Berg Balance Scale — The Berg Balance Scale is a clinical assessment tool used to measure an individual's ability to maintain balance during various functional tasks. The test includes 14 items, such as standing unsupported, reaching forward, turning, and standing on one leg. Each item is scored on a 5-point scale, ranging from 0 (unable to perform the task) to 4 (able to perform the task independently and safely). The scores for each item are summed to provide a total score, with a maximum possible score of 56.

SUMMARY:
This study aims to investigate the relationship between multifidus and gastrocnemius muscle thickness with postural stability in patients with spinal cord injury.

DETAILED DESCRIPTION:
Ultrasound imaging will be used to measure multifidus and gastrocnemius muscle thickness in patients with spinal cord injury. Postural stability will be assessed using the Berg Balance Scale, a clinical balance test consisting of 14 items that evaluate an individual's ability to maintain balance during various functional tasks such as standing unsupported, reaching forward, turning, and standing on one leg. The Berg Balance Scale is a reliable and valid clinical balance test that is commonly used in spinal cord injury patients. Statistical methods, including correlation and regression analysis, will be used to analyze the data and investigate the relationship between the multifidus and gastrocnemius muscle thickness and postural stability.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of spinal cord injury at least 6 months prior to study enrollment.
* Patients who are able to follow instructions and comply with study procedures.

Exclusion Criteria:

* Patients with severe cognitive impairment or inability to follow instructions.
* Patients with other medical conditions that may affect muscle thickness or postural stability, such as Parkinson's disease, multiple sclerosis, or severe osteoarthritis.
* Patients with contraindications for ultrasound imaging, such as pregnancy or implanted devices that may be affected by the imaging.
* Patients with severe motor deficits that may limit their ability to perform the study procedures.
* Patients who are unable to tolerate the testing procedures, such as the Berg Balance Scale or ultrasound imaging.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have spinal cord injury that gave consent to participate.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Relationship between multifidus thickness and postural stability | 1 day
  The relationship between multifidus muscle thickness measured by ultrasound in cm and results of berg scale will be measured statistically by calculating correlation coefficients.
  The Berg Balance Scale is a widely used clinical assessment tool designed to measure balance and stability in individuals who may have balance impairments due to various conditions such as stroke, Parkinson's disease, or multiple sclerosis. It consists of a series of 14 balance-related tasks that assess various aspects of balance, including sitting balance, standing balance, and dynamic balance.
  Each task is scored on a 5-point scale ranging from 0 to 4, with higher scores indicating better balance performance. The tasks involve different movements and challenges, such as maintaining sitting balance without arm support, standing up from a seated position, reaching forward while standing, turning around, and maintaining balance in different standing positions.
Relationship between gastrocnemius muscle thickness and postural stability | 1 day
  The relationship between gastrocnemius muscle thickness measured by ultrasound in cm and results of berg scale will be measured statistically by calculating correlation coefficients.
  The Berg Balance Scale is a widely used clinical assessment tool designed to measure balance and stability in individuals who may have balance impairments due to various conditions such as stroke, Parkinson's disease, or multiple sclerosis. It consists of a series of 14 balance-related tasks that assess various aspects of balance, including sitting balance, standing balance, and dynamic balance.
  Each task is scored on a 5-point scale ranging from 0 to 4, with higher scores indicating better balance performance. The tasks involve different movements and challenges, such as maintaining sitting balance without arm support, standing up from a seated position, reaching forward while standing, turning around, and maintaining balance in different standing positions.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa H Temel, M.D., Principal Investigator — Uskudar State Hospital

IPD SHARING:
Plan to Share IPD: Undecided
The individual participant data of this study will be shared upon reasonable request by corresponding author.